



## **ELM PARK, DUBLIN 4**

# Conway Institute of Bimolecular and Biomedical Research, University College Dublin, Belfield, Dublin 4

#### PARTICIPANT INFORMATION AND CONSENT FORM

STUDY TITLE: Food preference following Bariatric Surgery

#### NAME OF PRINCIPAL INVESTIGATOR:

Prof Carel le Roux MB MSc FRCP FRCPath PhD

## **Research Investigator**

Dr Loai Shakerdi

You are being invited to participate in a research study. Thank you for taking time to read this.

#### WHAT IS THE PURPOSE OF THIS STUDY?

Adults who are over weight and obese are at increased risk of developing associated health complications compared to patients who are of normal weight. An effective treatment of obesity is bariatric surgery. It has been shown to reduce blood pressure and improve diabetes in addition to its weight lowering effects. Among patients who have had bariatric surgery we see that their total food intake is reduced compared to before the operation. This will contribute to the weight loss as well. However we would like to understand more about why food intake changes by following up people over time that have undergone surgery and assessing their natural gut hormone response to food intake.

#### WHY HAVE I BEEN CHOSEN?

You have been chosen because you will be undergoing bariatric surgery.

Version 2 January 2016

WHAT WILL HAPPEN IF I VOLUNTEER?

Your participation is entirely voluntary. If you initially decide to take part you can

subsequently change your mind without difficulty. This will not affect your future

treatment in any way. Furthermore your doctor may decide to withdraw you from this

study if, he/she feels it is in your best interest.

If you agree to participate you will be invited to attend for a screening visit where any

questions you have will be addressed and you will be asked consent to the study. In

addition we will ask you to fill out a questionnaire regarding your food preferences.

The study will be conducted at the Clinical Research Centre at St Vincent's

University Hospital, Elm Park, Dublin 4.

There will be a total of **5 visits** to the research centre over a period of 2 years. On each

occasion you will be asked to attend having fasted from the night before. The visit

will commence at 10.30am. At each visit the research team conducting the study will

meet you. They will complete a questionnaire with you, complete measurements of

your weight, height and abdominal circumference. In addition you will have a blood

test, this will measure hormones produced by your gut that may be altered by surgery

and food. This will take 60-90 minutes to complete. Following this you will be

presented with a buffet meal containing foods of your liking and advised to eat until

you feel "comfortably full". Once again a blood test will be taken after the meal and

you are free to leave. The entire visit will take approximately 4 hours to complete.

The total amount of blood taken at each test is 10ml (approximately 1 tablespoons).

On two of the study visits an additional step is required. Before commencing the meal

you will be given an injection under the skin of a medication called Octreotide or

Saline (salty water). We would like to see the effect these treatments have on the

blood tests taken after your meal. Octreotide is a medication that is well-tolerated and

safe to use. Only one dose of Octreotide is required during the study. These visits will

take place at 12 months after your surgery.

The visits will take place 1 month prior to your operation, 3, 12 and 24 months after the surgery. At 12 months participants will be asked to attend on two occasions one

week apart for testing.

ARE THERE ANY BENEFITS FROM MY PARTICIPATION?

You will not directly benefit from participation in the study however the information

obtained from the study may help improve our understanding of the how bariatric

surgery in adult's works. This is not intended to replace routine medical assessments

with your GP or specialist.

ARE THERE ANY RISKS INVOLVED IN PARTICIPATING?

There may be some discomfort associated with blood sampling as the needle is

inserted into the vein. Sometimes there may be bruising after the blood sample is

taken and very rarely inflammation around the site of entry of the needle. Every

effort will be made to minimize risks. You will be monitored for any side effects to

the drug therapy given as part of the study.

You may feel some stinging or burning where we give the injection of saline (salty water)

and octreotide, but this usually only lasts a minute or so. We usually give these injections

beneath the skin on the abdomen or shoulder as it causes least discomfort.

Octreotide is a medication that resembles a natural hormone. It can be given as an

injection. It temporarily prevents release of other hormones from the gut after you have a

meal. It is commonly used in hospitals and considered a safe medicine. Some people

experience minor side effects such as nausea or abdominal discomfort after receiving this

injection, but if this happens it is usually transient. The medication is completely

eliminated from your body within about 8 hours, but some people may have loose bowel

motions the next day. Serious side effects are extremely rare, and the research team will

ask you about any medical problems that would make this medication unsafe for you to

take.

#### WHAT HAPPENS IF I DO NOT AGREE TO PARTICIPATE?

If you decide not to participate in this study your treatment will not be affected in any way.

#### **CONFIDENTIALITY**

Your identity will remain confidential. A study number will identify you. Your name will not be published or disclosed to anyone.

## **COMPENSATION**

Your doctors are adequately insured by virtue of their participation in the clinical indemnity scheme.

#### WHO IS ORGANISING AND FUNDING THIS RESEARCH?

This study is funded by a grant from the Health Research Board.

## WILL I BE PAID FOR TAKING PART IN THIS STUDY?

Participants will not be paid for participation in this study

# WILL MY EXPENSES BE COVERED FOR TAKING PART IN THIS STUDY?

Reasonable travel expenses will be reimbursed

#### HAS THIS STUDY BEEN REVIEWED BY AN ETHICS COMMITTEE?

The St. Vincent's Healthcare Group, Ethics and Medical Research Committee have reviewed and approved this study.

# **CONTACT DETAILS**

Dr Loai Shakerdi

Conway Institute of biomolecular and biomedical research

University College Dublin

Belfield

Dublin4

Phone: 089 2214185

Email: guthormonestudy@gmail.com

# PLEASE TICK YOUR RESPONSE IN THE APPROPRIATE BOX

| • | I have read and understood the Participant Information | YES □ NO □ |
|---|---|---|
| • | I have had the opportunity to ask questions and discuss the study | YES □ NO □ |
| • | I have received satisfactory answers to all my questions | YES $\square$ NO $\square$ |
| • | I have received enough information about this study | YES $\square$ NO $\square$ |
| • | I understand that I am free to withdraw from the study at any time without giving a reason and without this affecting my future medical care I agree to take part in the study | YES NO YES NO |
| Participant's Signature: | | Date: |
| Participant's Name in print: | | |
| Investigator's Signature: | | Date: |
| Investigator's Name in print: | | _ |